CLINICAL TRIAL: NCT04930614
Title: Prevalence and Associated Risk Factors of HIV Infections in a Representative Transgender and Non-binary Population in Flanders and Brussels (Belgium): A Community-based, Cross-sectional Study Using Time-location Sampling
Brief Title: Prevalence and Risk Factors of HIV Infections in Transgender and Non-binary People in Flanders and Brussels (Belgium)
Status: Completed | Type: Observational
Sponsor: Centre for Evidence-Based Practice, Belgium (Other)
Collaborators: University Hospital, Ghent (Other); Institute of Tropical Medicine, Belgium (Other); Institute for the Equality of Women and Men, Belgium (Unknown); Gilead Sciences (Industry); Belgian Red Cross (Other)
Responsible Party: Sponsor
Other Study IDs: HIV-001
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
Keywords: HIV; Transgender and non-binary people; LGBT+; time-location sampling; risk factor
MeSH Terms: conditions — HIV Infections | interventions — Sex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Oral fluid aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender and non-binary people: Adult transgender and non-binary people in Flanders and Brussels (Belgium)
  Interventions: Other: Survey on socio-demographic variables and healthcare-seeking, sexual and drug-using behaviour

INTERVENTIONS:
Other: Survey on socio-demographic variables and healthcare-seeking, sexual and drug-using behaviour — Digital survey to estimate the associated risk factors for HIV infections in transgender and non-binary people in Flanders and Brussels (Belgium)

SUMMARY:
Background: HIV prevalence and sexual risk have been estimated very high for transgender people. However, the limited sampling and data collection methods used in current research on transgender people potentially led to overrepresentation and generalisation of people at risk for HIV. Current HIV prevalence estimates in transgender populations are generalised from studies mainly focusing on transgender women who engage in sex work. Moreover, current research remains cisnormative, and studies focusing on non-binary people, who identify with a broad range of identities beyond the traditional male and female gender identities, are scarce.

Objective: This study aims to estimate the HIV prevalence rate in the Flemish and Brussels (Belgium) transgender population, including transgender women as well as transgender men and non-binary people, and identifying the associated individual and community-level risk factors.

Methods: In this community-based cross-sectional study, self-identified transgender and non-binary (TGNB) people will be recruited through a two-stage time-location sampling approach to minimize selection bias. In a first part, community settings in which TGNB people gather will be mapped using qualitative and ethnographic research methods, to reveal how the TGNB community in Flanders and Brussels is structured and to develop an accurate sampling frame. In a second part, to select the respondents, a multistage sampling design is applied involving a stratification based on setting type (healthcare facilities vs outreach events), a selection of clusters by systematic sampling and a simple random selection of TGNB people within each cluster. Participants will complete an electronic self-reported survey to measure sociological, sexual and drug-using behaviors (risk factors) and, at the same time, oral fluid aliquots will be collected and tested for HIV antibodies. Logistic regression models will be used to evaluate risk factors independently associated with HIV infection.

Conclusion: To the best of our knowledge, this study will be the first to investigate the HIV prevalence rates and behaviors that increase risk and vulnerability for HIV infection in an accurate representation of the TGNB population in a West European country. The findings of this study will globally serve as a knowledge base for identifying subgroups at risk for becoming infected with HIV within TGNB people and to set up targeted prevention programs on sexual health.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) self-identified transgender and non-binary people
* Able to read, write and understand the survey
* Consent to participate in the survey and to self-collect an oral fluid sample

Exclusion Criteria:

* Cisgender people
* People who have no understanding of the multilingual survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women and transgender men, as well as non-binary people are included in this study. Transvestite or crossdressing people who identify as transgender are also included.
Study Population: The study population involves transgender (identifying more with the opposite gender than the gender which was assigned at birth) and non-binary (identifying with both or neither binary genders) people in Flanders and Brussels.
Sampling Method: Probability Sample
Enrollment: 1068 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
HIV infection | Study duration (one year)
  Oral fluid samples will be self-collected by the participants through swabbing and tested for the presence of HIV antibodies with the DPP HIV1/2 Assay (Chembio Diagnostic Systems, Inc) at the Institute of Tropical Medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Guy T'Sjoen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Brier N, Van Schuylenbergh J, Van Remoortel H, Van den Bossche D, Fieuws S, Molenberghs G, De Buck E, T'Sjoen G, Compernolle V, Platteau T, Motmans J. Prevalence and associated risk factors of HIV infections in a representative transgender and non-binary population in Flanders and Brussels (Belgium): Protocol for a community-based, cross-sectional study using time-location sampling. PLoS One. 2022 Apr 11;17(4):e0266078. doi: 10.1371/journal.pone.0266078. eCollection 2022. PMID 35404977